CLINICAL TRIAL: NCT04898790
Title: Promoting Physical Activity to Improve Cognitive Function in Older Adults Undergoing Hematopoietic Cell Transplantation
Brief Title: Improving Cognitive Function in Older Adults Undergoing Stem Cell Transplant
Acronym: PROACTIVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0421-21-EP
Record Dates: First submitted 2021-05-07; First posted 2021-05-24 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Leukemia; Lymphoma; Multiple Myeloma; Myelodysplastic Syndromes (MDS); Myeloproliferative Neoplasm
Keywords: Hematopoietic cell transplantation
MeSH Terms: conditions — Leukemia; Lymphoma; Multiple Myeloma; Myelodysplastic Syndromes; Myeloproliferative Disorders

STUDY DESIGN:
Intervention Model Description: Aim 1 will seek feedback from 1)adult participants 60+ years who have recently undergone HCT, 2)participants' care-partner, and 3)HCT team members for preliminary adaptation of the evidence-based physical activity intervention (CHAMPS-II) manual, and development of study materials.
  Aim 2 will iteratively adapt and implement CHAMPS-II for adults 60 years and older undergoing HCT with feedback from 1)adult participants 60+ years receiving HCT, 2)participants' care-partner, and 3)HCT team members.
  Aim 3 will take the final CHAMPS-II adaptation from Aim 2 and pilot test it, using a Type 1 hybrid effectiveness-implementation design to determine its preliminary effectiveness to improve cognitive function compared to a wait-list control condition. Feedback will be obtained on the intervention and control condition from 1)adult participants 60+ years receiving HCT, 2)participants' care-partner, and 3)HCT team members.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor completing primary outcome testing during the RCT in Aim 3 will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Feedback for Preliminary Adaptation (No Intervention): Participants in Aim 1 will participate in qualitative interviews to obtain feedback on the CHAMPS-II intervention and survivorship education active control condition materials. Interviews will be with 1)adult participants 60+ years who have recently undergone HCT, 2)participants' care-partner, and 3)HCT team members.
- Adapted CHAMPS-II intervention (Experimental): All participants in Aim 2 (preliminary testing) and Aim 3 (RCT) will participate in the CHAMPS-II physical activity program adapted to the HCT setting. Testing for outcome measures will be completed, and feedback on the intervention will be obtained via qualitative interviews from 1)adult participants 60+ years receiving HCT, 2)participants' care-partner, and 3)HCT team members.
  Aim 3 participants will be randomized to either the immediate intervention (intervention then follow-up) or delayed intervention (wait period and then intervention).
  Interventions: Behavioral: CHAMPS-II adapted to adults 60+ years in HCT setting

INTERVENTIONS:
Behavioral: CHAMPS-II adapted to adults 60+ years in HCT setting — CHAMPS-II is an evidence-based physical activity program designed to increase physical activity in sedentary older adults with multiple chronic health conditions. This is an individually tailored program that provides information, skills, training, and problem-solving support to older adults. Participants will engage in progressive, light to moderate-intensity physical activity throughout the HCT process, with the support of physical therapists, physical activity counselors, and their care-partner. They will take part in supervised exercise sessions; unsupervised exercise sessions; counseling sessions to address barriers, motivators, goals, and safety; and receive telephone support. Walking is the primary mode of aerobic activity, with training in flexibility, strengthening and balance exercises also included. An exercise kit will be provided, consisting of an intervention workbook, therapeutic resistance bands, and activity logs.
  Arms: Adapted CHAMPS-II intervention

SUMMARY:
Cancer and treatment-related cognitive changes, such as thinking or remembering, hinder resumption of normal routine and roles and worsen quality of life. Older adults undergoing hematopoietic cell transplantation (HCT) are at high-risk for cognitive impairment. Age is a risk factor for Alzheimer's Dementia (AD) and the hematological malignancies leading to HCT. There are shared mechanisms and interactions between AD and cancer-related cognitive decline (CRCD). Physical activity improves cognitive function in older adults and survivors of other cancers. This study hypothesizes that increasing physical activity can also improve cognitive function in this vulnerable population.

The study has two goals. The first is to adapt and test an evidence-based physical activity intervention, The Community Health Activities Model Program for Seniors II (CHAMPS II), in the HCT setting for adults 55 years and older. This will be done using semi-structured interview of up to 10 patients who have experienced the HCT process within the last 3 to 6 months with HCT care-team partners.

The second goal will explore the prevalence and impact of AD-neuropathology and inflammation on cancer-related cognitive decline (CRCD) in older adults undergoing HCT.

DETAILED DESCRIPTION:
Hematologic malignancies are diseases that primarily affect older adults, with a median age at diagnosis of 65 years. Hematopoietic cell transplantation (HCT) is a potentially curative and life-prolonging treatment for patients with hematologic malignancies. Cancer and treatment-related cognitive changes cause distress, hinder resumption of normal routine and roles, and worsen quality of life. HCT differs from the delivery of chemotherapy in other cancer settings due to the intensity of chemotherapy and severity of toxicity. Older adults undergoing HCT are at high risk for cognitive decline and pervasive cognitive deficits. Interventions to improve cognitive outcomes are needed. The prevalence and risk of cognitive decline post-HCT are greater for older adults because of a greater number of existing health conditions (i.e., vascular disease) and impaired physical and psychologic function pre-HCT that can be exacerbated by treatment and the overall HCT experience.

Exercise training improves cancer-related health outcomes, including cardiorespiratory fitness, inflammation, cancer related fatigue, depressive symptoms, and sleep disturbance. There is consistent evidence showing that physical activity improves cognitive function in older adults and survivors of other cancers. Improvement in cardiorespiratory fitness, brain structure, and inflammation underlie the mechanisms of the cognitive benefits of physical activity. While untested in older adults undergoing HCT, the investigator hypothesizes that increasing physical activity can also improve cognitive function in this vulnerable population.

Physical activity improves the cognitive domains most affected by cancer treatment, namely executive function and working memory. Cognitive function is an important outcome to older adults and has not been a focus of physical activity interventions in the HCT population. In addition, older adults are underrepresented in previous physical activity interventions in the HCT population.

Investigators will adapt CHAMPS II, an evidence-based physical activity intervention, to the HCT setting for older adults to improve cognitive function. This is an individually tailored program that provides information, skills, training, and problem-solving support to older adults. The program provides a foundation for application by including an instructor manual and directions for implementation. CHAMPS-II has been adapted and implemented in diverse communities using existing resources and improving contextual factors to increase physical activity for sedentary older adults.

Adaptation of evidence-based interventions, such as CHAMPS-II, can result in an attenuation of effects if the core components are not maintained. However, adaptations can be made to fit the needs and priorities of the service setting, target audience, mode of delivery, and cultural context without compromising CHAMPS-II effectiveness. Through a research-practice partnership approach, investigators will help adapt the program while maintaining the core components of CHAMPS-II, develop new program materials, provide training, monitor implementation, and conduct program evaluation. The overarching goal is to enable HCT team members to implement CHAMPS-II and leverage existing organizational resources to enhance feasibility and sustainability.

The research plan proposes a hybrid effectiveness-implementation design, which is a design that spans the effectiveness and implementation research to accelerate the translation of physical activity interventions into practice for older adults with cancer. This novel trial design will allow testing of the program within a randomized clinical trial methodology while observing and gathering information on implementation. The effectiveness study condition offers an ideal opportunity to examine implementation issues and plan for implementation strategies for a future study that examines both effectiveness and implementation strategies. The study will use the RE-AIM (Reach, Effectiveness - Adoption, Implementation, and Maintenance) framework for planning and formative and process evaluation of the intervention. Formative and process evaluation provides information needed to evaluate an intervention's potential for translation into clinical practice.

Investigators aim to understand the prevalence and impact of AD-neuropathology and inflammation on cognitive function and structural brain changes in older adults undergoing HCT. Quantifiable AD-related neuropathology can accumulate silently for decades with no clinical symptoms. Some will have no AD pathology, some will have "silent" AD pathology, and some will have clinically relevant levels of AD pathology. Brain volumes is also a measure of cognitive reserve with many factors that could impact brain volumes including aging, AD, other degenerative diseases, untreated obstructive sleep apnea (OSA), chronic stress, and ethyl alcohol or ethanol abuse (ETOH). Some patients with low brain volumes may have negative AD biomarkers. However, brain volumes may be a good predictor of CRCD. Investigators expect to gain an understanding of the prevalence of between-subject variability in the quantity of AD neuropathology and differences in brain volume. The results of this research will lay the groundwork for future funding opportunities to elucidate the bidirectional mechanisms, prevention and treatment of AD and CRCD in this population.

ELIGIBILITY:
Arm 1:

Inclusion Criteria for Participants:

* age 60 years and older
* have a diagnosis of hematological malignancy
* have received autologous or allogeneic HCT within the prior 3-6 months
* able to speak and read English
* have provided written informed consent

Exclusion Criteria for Participants:

* there are no exclusion criteria

Inclusion Criteria for Participants' Care-Partner:

* age 19 years and older
* able to speak and read English

Exclusion Criteria for Participants' Care-Partner:

* there are no exclusion criteria

Inclusion Criteria for Transplant Team Member:

* age 19 years and older
* able to speak and read English

Exclusion Criteria for Transplant Team Member:

* there are no exclusion criteria

Arms 2 and 3:

Inclusion Criteria for Participants:

* age 55 years and older
* have a diagnosis of hematological malignancy
* planned to receive an autologous or allogeneic HCT
* able to walk 4 meters as part of the Short Physical Performance Battery (with or without assistance)
* (In Arm 3 only): willingness to be randomized to either initiate the physical activity intervention pre-HCT or following Day 180 post-HCT, and to follow the protocol for the group to which they have been assigned
* able to speak and read English
* have provided written informed consent

Exclusion Criteria for Participants:

* development of chest pain, severe shortness of breath, or occurrence of other safety concerns during the physical performance measures (i.e. Short Physical Performance Battery)
* is not cleared to participate in exercise by a physician

Individuals with the following current conditions/diagnoses documented in medical history will be required to provide clearance for exercise from their cardiologist:

* Myocardial infarctions in the past 3 months
* Resting or unstable angina
* Uncontrolled and/or serious arrhythmias
* 3rd degree heart block
* Acute congestive heart failure or ejection fraction <30%
* Clinically significant aortic stenosis

Individuals with the following conditions/diagnoses will be required to provide clearance for exercise from their surgeon:

* Hip fracture, hip or knee replacement, or spinal surgery in the past 3 months

  * other medical, psychiatric, or behavioral factors that in the judgement of the principal investigator may interfere with study participation or the ability to follow either the intervention or the active control condition
  * (In Arm 3 for those who agree to the voluntary measures of blood, saliva and MRI, there are additional exclusions to avoid conditions that may confound study outcomes):
* history of residual brain abnormalities from prior severe traumatic brain injury (e.g. encephalomalacia) or other significant abnormalities documented on a recent brain MRI (e.g. brain cancer, large vessel strokes, residual subdural hematoma)
* history of major stroke with obvious residual deficits
* history of relapsing and remitting Multiple Sclerosis
* active moderate to severe psychiatric symptoms due to primary psychiatric disorder

Inclusion Criteria for Participants' Care-Partner:

* age 19 years and older
* able to speak and read English
* able to walk 4 meters as part of the Short Physical Performance Battery (with or without assistance)
* have no medical contraindications for participating in light to moderate-intensity physical activity per PI review of medical history as reported on the care-partner medical history form

Exclusion Criteria for Participants' Care-Partner:

* development of chest pain, severe shortness of breath, or occurrence of other safety concerns during the physical performance measures (i.e. Short Physical Performance Battery)
* is not cleared to participate in exercise by a physician

Individuals with the following current conditions/diagnoses documented in medical history will be required to provide clearance for exercise from their cardiologist:

* Myocardial infarctions in the past 3 months
* Resting or unstable angina
* Uncontrolled and/or serious arrhythmias
* 3rd degree heart block
* Acute congestive heart failure or ejection fraction <30%
* Clinically significant aortic stenosis

Individuals with the following conditions/diagnoses will be required to provide clearance for exercise from their surgeon:

o Hip fracture, hip or knee replacement, or spinal surgery in the past 3 months

* other medical, psychiatric, or behavioral factors that in the judgement of the principal investigator may interfere with study participation or the ability to follow either the intervention or the active control condition

Inclusion Criteria for Transplant Team Member:

* age 19 years and older
* able to speak and read English

Exclusion Criteria for Transplant Team Member:

* there are no exclusion criteria

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2021-11-18 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Change in executive function as measured by Trails A. | 12 weeks
  Change in raw scores and z-scores, determined by the following neuropsychological test: Trail Making Test Part A (Trails A). Time to complete and number of errors are measured, where less time and errors are better outcomes.
Change in executive function as measured by Trails B. | 12 weeks
  Change in raw scores and z-scores, determined by the following neuropsychological tests: Trail Making Test Part B (Trails B). Time to complete and number of errors are measured, where less time and errors are better outcomes.
Change in executive function as measured by the Controlled Oral Word Association Test (COWAT). | 12 weeks
  Change in raw scores and z-scores, determined by the following neuropsychological test: Controlled Oral Word Association Test (COWAT). Minimum score is zero and maximum is unlimited; higher score means better outcome.
Change in working memory as measured by the Hopkins Verbal Learning Test-Revised (HVLT-R). | 12 weeks
  Change in raw scores and z-scores, determined by the following neuropsychological test: Hopkins Verbal Learning Test-Revised (HVLT-R). There are 3 learning trials and 1 delayed recall trial. Minimum score for each is zero and maximum is 12; higher score means better outcome. There is also a delayed recognition trial where person is presented with both true positives and false positives. Minimum score for both is zero and maximum is 12. For the true positives a higher score means better outcome. For the false positives a lower score means better outcome.

SECONDARY OUTCOMES:
Change in global cognitive function as measured by the Montreal Cognitive Assessment (MoCA). | 12 weeks
  Change in total score, determined by objective measures of global cognitive function using the Montreal Cognitive Assessment (MoCA). Minimum score is zero and maximum is 30; higher score means better outcome.
Change in subjective memory as measured by the Neuro-Quality of Life (QOL) Cognition Function-Short Form. | 12 weeks
  Change in total score, determined by patient questionnaire: Neuro-Quality of Life (QOL) Cognition Function-Short Form. Minimum score is 8 and maximum score is 40; higher score means better outcome.

OTHER OUTCOMES:
Change in functional ability as measured by the Short Performance Physical Battery (SPPB). | 12 weeks
  Change in total score, determined by objective measures of balance, gait speed and endurance with the Short Performance Physical Battery (SPPB). Minimum score is zero, maximum is 12; higher score means better outcome.
Change in endurance as measured by the 6-minute walk. | 12 weeks
  Change in distance measured in meters, determined by a 6-minute walk. More distance in meters is better outcome.
Change in performance of instrumental activities of daily living as measured by the Lawton Instrumental Activities of Daily Living (IADL). | 12 weeks
  Change in total score, determined by a self-report questionnaire: Lawton Instrumental Activities of Daily Living (Lawton IADL). Minimum score is zero, maximum is 8; higher score means better outcome.
Change in physical activity as measured by the Community Healthy Activities Model Program for Seniors II (CHAMPS-II) questionnaire. | 12 weeks
  Change in total score of light and moderate physical activity as measured by a self-report questionnaire (CHAMPS-II questionnaire). Frequency and duration of various intensity activities and their caloric expenditure per week are all scored. No activity, duration or calories expended would be minimum score, and unlimited would be the maximum; where more frequency, duration and calories expended would be a better outcome.
Change in physical activity as measured by the activPAL4 accelerometer data. | 12 weeks
  Change in time spent in upright postural allocation as measured by an accelerometer (activPAL4). Increased time in upright postural allocation is better outcome.
Change in brain volume as measured by MRI brain. | 52 weeks
  The focal measures collected for this study include structural atrophy of the hippocampus and cortical thickness of neocortical regions reflecting neurodegeneration (AD-related atrophy), as assessed with high-resolution anatomical MRI.
Change in AD biomarkers as measured by plasma Tau and p-Tau 217. | 52 weeks
  The characteristic neurofibrillary tangles of AD are composed of pathological tau proteins. Two different measures of tau will be obtained: total tau and phosphorylated tau 217 (p Tau-217). Total tau will be assayed with a Quanterix Simoa Tau 2.1 Kit. The design of this assay identifies all isoforms of the tau protein, hence "total tau". Phosphorylated tau-217 (p-Tau 217) will be assayed with a Quanterix ALZPath Simoa p-Tau217 V2 Assay Service.
Change in biomarkers of inflammation as measured by IL6, IL8, IL10, TNF alpha, and CRP. | 52 weeks
  Quanterix will measure IL-6, IL-8, IL-10 and TNFa via a Kit Hu 4-Plex SP-116 for cytokines, and C-reactive protein (CRP) via a Simoa CRP Developer Kit.
Presence or absence of AD-related neuropathology as measured by APOE e4 carrier status. | Baseline pre-HCT
  AD genotyping for APOE alleles will be collected via a saliva swab. Apolipoprotein E (APOE) is a complex glycolipoprotein that facilitates the uptake, transport, and distribution of lipids. Numerous studies have shown cognitive vulnerability in non-demented APOE-e4 carriers relative to non-APOE-e4 carriers. APOE will be processed by Salimetrix.

CONTACTS AND LOCATIONS:
Overall Officials: Thuy Koll, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No